CLINICAL TRIAL: NCT00925431
Title: Lifestyle Modification Program for Overweight and Obese Fibromyalgia Patients
Brief Title: Nutrition and Coping Education for Symptom and Weight Management for Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Akiko Okifuji, PhD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21744; R21AR055114 (NIH)
Record Dates: First submitted 2009-06-18; First posted 2009-06-22 (Estimated); Last update posted 2023-07-24 (Actual); Status verified 2017-03

CONDITIONS: Fibromyalgia; Obesity
MeSH Terms: conditions — Fibromyalgia; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle Modification (Experimental): Behavioral: cognitive-motivational enhancement to lifestyle management plus nutritional education.
  Interventions: Behavioral: Lifestyle Modification
- Supportive education (Active Comparator): General fibromyalgia education plus nutritional education.
  Interventions: Behavioral: Supportive education

INTERVENTIONS:
Behavioral: Lifestyle Modification — 16 hours of motivational, lifestyle management session, 8 hours nutritional education.
  Arms: Lifestyle Modification
Behavioral: Supportive education — 16 hours general fibromyalgia education, 8 hours of nutritional education
  Arms: Supportive education

SUMMARY:
Research has shown that weight problems are very common in fibromyalgia. Research also suggests that overweight and obesity may contribute to worsening of fibromyalgia symptoms and biochemical vulnerability associated with fibromyalgia. Effective weight management may be important in not only improving general health but also better management of fibromyalgia symptoms. Research has indicated that nutrition and coping education is important aspects of successful weight management. In this study, the investigators are evaluating the effect of nutrition and coping education on weight and symptom management of fibromyalgia among overweight and obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia patients whose body mass index is greater than 25.
* Age 21-65 of both sex and all race.

Exclusion Criteria:

* Co-occurring progressive disease
* Planning to have surgery in the next year
* Pregnancy or planning to be pregnant in the next year
* Having known cardiovascular diseases
* Having known serious psychopathology (Diagnoses of psychosis, organic mental disorder, dissociative disorder, active suicidal intent, inpatient admission to psychiatric ward in the past year, evidence of self-injurious behaviors in the past year, current or recent history (2years) of non-IV substance abuse, any history of recreational IV drug use)
* Having autoimmune disorder (e.g., rheumatoid arthritis)
* Having neuropathic pain
* Having pain associated with terminal illness, acute pain, pain associated with specific organ damage (eg, stomach ulcer)
* Concurrent use of weight controlling medications (eg, Xenical)
* A history of weight reduction surgery
* Concurrent participation in weight loss programs or other cognitive-behavioral coping therapy
* Self-reported physician diagnosed conditions of chronic bronchitis, asthma, or emphysema
* Report history of head injury, neurological illness, diagnosis of learning disability, learning problems, or special education, substantial toxin or chemical exposure within five years of FMS onset, near drowning, recreational IV drug use

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Major FM syndrome symptoms and weight changes | Pre-treatment, Post-treatment, 3 follow-ups

SECONDARY OUTCOMES:
Obesity-related health quality of life | Pre-treatment, Post-treatment, 3 month FU
FMS-related neuroendocrine factors and obesity-related health indices | Pre-treatment, post-treatment, 3 month FU

CONTACTS AND LOCATIONS:
Overall Officials: Akiko Okifuji, PhD, Principal Investigator — University of Utah
Locations (1):
- Pain Research Center, University of Utah, Salt Lake City, Utah, United States